CLINICAL TRIAL: NCT01860859
Title: Randomized Controlled Trial Comparing Three Techniques of Uterine Closure on the Myometrium Thickness Evaluated With Ultrasound Six Months After a Primary Cesarean
Brief Title: Suture of UTerus and Ultrasound Repair Evaluation
Acronym: SUTURE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Laval University (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Emmanuel Bujold, MD, MSc, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: C12-03-204
Record Dates: First submitted 2013-05-09; First posted 2013-05-23 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Uterine Scar Defect
Keywords: cesarean; ultrasound; hysterotomy; uterus; suture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Unlocked double layer (Other): Double layer closure with a first continuous unlocked suture of the deep portion of the myometrium avoiding the inclusion of the decidua and a second unlocked continuous suture that approximate the upper portion of the myometrium.
  Interventions: Procedure: Closure of the hysterotomy at the time of primary cesarean
- Locked single layer closure (Other): As reported in Williams Obstetrics textbook
  Interventions: Procedure: Closure of the hysterotomy at the time of primary cesarean
- Locked double layer (Other): Double layer closure with a first continuous locked suture and a second imbricating continuous suture.
  Interventions: Procedure: Closure of the hysterotomy at the time of primary cesarean

INTERVENTIONS:
Procedure: Closure of the hysterotomy at the time of primary cesarean

SUMMARY:
This study compares three techniques of uterine closure on myometrium thickness evaluated by ultrasound six months after the primary cesarean. The three techniques include: 1) locked single layer closure; 2) double layer closure with a first continuous locked suture and a second imbricating continuous suture; 3) double layer closure with a first continuous unlocked suture of the deep portion of the myometrium avoiding the inclusion of the decidua and a second unlocked continuous suture that approximate the upper portion of the myometrium. The primary outcome is the mean myometrium thickness at the site of the uterine scar evaluated by transvaginal ultrasound at six months after cesarean.

ELIGIBILITY:
Inclusion Criteria:

* Planned cesarean
* Primary cesarean
* ≥ 38 gestational weeks

Exclusion Criteria:

* Previous cesarean
* Women < 18 years old
* Multiple gestation
* Mullerian anomalies
* Active labor
* Diabetes
* BMI >35 kg/m2
* Placenta praevia
* Chronic systemic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Mean myometrium thickness | 6 months after intervention
  Using transvaginal ultrasound the residual myometrium thickness at the site of the uterine scar will be measure.

SECONDARY OUTCOMES:
Estimated blood loss | Same day of intervention: day 1
Operative time | Same day of intervention: day 1
Mean number of haemostatic sutures | Same day of intervention: day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Québec, Québec, Quebec, Canada

REFERENCES:
- [Background] Roberge S, Boutin A, Chaillet N, Moore L, Jastrow N, Demers S, Bujold E. Systematic review of cesarean scar assessment in the nonpregnant state: imaging techniques and uterine scar defect. Am J Perinatol. 2012 Jun;29(6):465-71. doi: 10.1055/s-0032-1304829. Epub 2012 Mar 7. PMID 22399223
- [Background] Roberge S, Chaillet N, Boutin A, Moore L, Jastrow N, Brassard N, Gauthier RJ, Hudic I, Shipp TD, Weimar CH, Fatusic Z, Demers S, Bujold E. Single- versus double-layer closure of the hysterotomy incision during cesarean delivery and risk of uterine rupture. Int J Gynaecol Obstet. 2011 Oct;115(1):5-10. doi: 10.1016/j.ijgo.2011.04.013. Epub 2011 Jul 26. PMID 21794864